CLINICAL TRIAL: NCT06078657
Title: Prospective, Single-arm Phase II Exploratory Study of the Efficacy and Safety of IBI110 Combined With Sintilimab in Advanced or Metastatic Esophageal Squamous Cell Carcinoma That Has Failed First-line Anti-PD-1 Antibody Therapy
Brief Title: IBI110 Combined With Sintilimab in Second-line Advanced or Metastatic Esophageal Squamous Cell Carcinoma(ESCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Doctor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI110Y006
Record Dates: First submitted 2023-09-21; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC); PD-1 Inhibitors
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI110 combined with Sintilimab (Experimental)
  Interventions: Drug: IBI110+Sintilimab

INTERVENTIONS:
Drug: IBI110+Sintilimab — IBI110, 200mg, intravenously on the first day of each cycle, every 3 weeks for 1 cycle (Q3W), and the maximum use time was 2 years.
  Sintilimab, 200mg, intravenously on the first day of each cycle, every 3 weeks as a cycle (Q3W), and the maximum use time was 2 years.

SUMMARY:
This is a single-center, prospective, single-arm Phase II clinical study to evaluate the efficacy and safety of IBI110 in combination with Sintilimab in subjects with advanced or metastatic esophageal squamous cell carcinoma (ESCC) who have failed first-line treatment with PD-1 inhibitors combined with chemotherapy.

Patients who meet the inclusion criteria will be treated with IBI110 combined with Sintilimab until disease progression, death, toxicity intolerance, withdrawal of informed consent, initiation of new anti-tumor therapy, or termination of therapy for other reasons specified in the protocol. RECIST v1.1 was used for clinical tumor imaging evaluation every 6 weeks during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent prior to the implementation of any procedures related to the trial, and be able to comply with protocol visits and related procedures;
* Age ≥18 years old and ≤75 years old;
* Unresectable, locally advanced recurrent or metastatic esophageal squamous cell carcinoma confirmed by histopathological examination (excluding adenosquamous cell carcinoma mixed type and other pathological types);
* Disease progression must have previously received first-line anti-PD-1 antibody combined with chemotherapy, and disease progression must occur after at least 2 imaging evaluations after anti-PD-1 therapy (the second imaging evaluation is not less than 84 days after the first anti-PD-1 therapy); And the best efficacy evaluation of CR or PR population; It takes ≥6 months for the disease to stabilize in SD population.
* First-line chemotherapy includes fluorouracil combined with cisplatin or paclitaxel combined with cisplatin;
* Did not receive any systematic therapy, such as chemotherapy, targeted therapy, immunotherapy or other therapy, for 21 days before enrollment;
* Occurrence of immune-related adverse events during prior treatment with anti-PD-1 antibodies, except for the following: a.Grade 3 or higher immune-related adverse events (ir-AE) occurred, except for asymptomatic non-bullous or non-exfoliating rashes;b.did not recover from grade 2 immune-related adverse events (ir-AE);c.any adverse events leading to permanent discontinuation of PD-1;
* Note: Any level of toxicity that requires replacement therapy and is stable (such as thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is permissible.
* There was at least one radiographically measurable lesion according to the solid tumor efficacy evaluation criteria (RECIST v1.1 edition).
* ECOG score 0-1;
* Expected survival time >3 months;
* For adequate organ function, the subject must meet the following laboratory criteria:

  1. The absolute value of neutrophil (ANC) ≥1.5x109/L in the past 14 days without the use of granulocyte colony-stimulating factor;
  2. Platelets ≥100×109/L without blood transfusion in the past 14 days;
  3. Hemoglobin >9g/dL in the last 14 days without blood transfusion or use of erythropoietin;
  4. Total bilirubin ≤1.5× upper limit of normal (ULN);
  5. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN (ALT or AST ≤5×ULN for subjects with liver metastasis);
  6. Serum creatinine ≤1.5×ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 ml/min;
  7. Good coagulation function, defined as International standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
  8. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
  9. The myocardial enzyme profile was within the normal range (if the researcher comprehensively judged that the simple laboratory abnormality was not clinically significant, it was also allowed to be included);
* For female subjects of reproductive age, a urine or serum pregnancy test should be performed negative within 3 days prior to receiving the first study drug administration (day 1 of cycle 1). If the urine pregnancy test results cannot be confirmed as negative, a blood pregnancy test is requested. Women of non-reproductive age were defined as at least one year after menopause or having undergone surgical sterilization or hysterectomy;
* If there is a risk of conception, all subjects (male or female) are required to use a contraceptive with an annual failure rate of less than 1% for the entire duration of treatment up to 120 days after the last study drug administration (or 180 days after the last study drug administration).

Exclusion Criteria:

* Esophageal squamous cell carcinoma known to be prone to complete obstruction under endoscopy requires interventional therapy to relieve the obstruction;
* After stent implantation in esophagus or trachea; Patients who are at high risk of bleeding or perforation due to significant tumor invasion of adjacent organs (aorta or trachea), or who have developed fistulas;
* Malignant diseases other than esophageal cancer diagnosed within 3 years prior to initial administration (excluding radical basal cell carcinoma of the skin, squamous epithelial carcinoma of the skin, and/or carcinoma in situ after radical resection);
* An active autoimmune disease requiring systemic treatment (e.g. with disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred within 2 years prior to initial administration. Replacement therapies (such as thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy;
* Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* Allergy to Sintilimab, IBI110 active ingredients or excipients of this study is known;
* Prior treatment with anti-LAG-3 antibodies;
* Has not fully recovered from toxicity and/or complications caused by any intervention before starting treatment (i.e., ≤ grade 1 or baseline, excluding weakness or hair loss);
* Received the following treatment:

  1. Received systemic anti-tumor therapy within 3 weeks before treatment, such as chemotherapy, targeted therapy, immunotherapy (including Chinese herbal therapy with anti-tumor indications), etc.;
  2. Received any investigational drug therapy within 4 weeks prior to treatment;
  3. Receiving excessive doses of immunosuppressive drugs (systemic corticosteroids exceeding 10mg/ day of prednisone or its equivalent) within 4 weeks prior to treatment;
  4. Received live attenuated vaccine within 4 weeks prior to treatment (or plan to receive live attenuated vaccine during the study period);
  5. Major surgery, or unhealed surgical wounds, ulcers, or fractures within 4 weeks prior to treatment.
* An active autoimmune disease requiring systemic treatment (e.g. with disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred within 2 years prior to first administration. Replacement therapies (such as thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy;
* Known allogeneic organ transplantation (other than corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* People who are known to be allergic to the active ingredient or excipient of Sintilimab in this study;
* Has not fully recovered from toxicity and/or complications caused by any intervention before starting treatment (i.e., ≤ grade 1 or baseline, excluding weakness or hair loss);
* Known history of human immunodeficiency virus (HIV) infection (i.e., HIV1/2 antibody positive);
* Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected greater than the upper limit of normal value in the laboratory of the study center);
* Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

  1. HBV viral load <1000 copies /ml (200IU/ml) prior to initial administration, subjects should receive anti-HBV therapy throughout the study chemotherapy drug treatment to avoid viral reactivation
  2. For subjects with anti-HBC (+), HBsAg (-), anti-HBS (-) and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of viral reactivation is required
* Active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection);
* Pregnant or lactating women;
* The presence of any serious or uncontrolled systemic disease, such as:

  1. The resting electrocardiogram has major abnormal rhythm, conduction or morphology, such as complete left bundle branch block, heart block above Ⅱ degree, ventricular arrhythmia or atrial fibrillation;
  2. Unstable angina pectoris, congestive heart failure, New York Heart Association (NYHA) grade ≥2 chronic heart failure;
  3. Any arterial thrombosis, embolism or ischemia occurred within 6 months before treatment, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack;
  4. Poor blood pressure control (systolic > 140mmHg, diastolic > 90mmHg);
  5. There is a history of non-infectious pneumonia requiring glucocorticoid therapy within 1 year prior to first administration, or there is currently clinically active interstitial lung disease;
  6. Active pulmonary tuberculosis;
  7. There is an active or uncontrolled infection that requires systemic treatment;
  8. Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;
  9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
  10. Poor diabetes control (fasting blood glucose (FBG) > 10mmol/L);
  11. Urine routine indicated urine protein ≥++, and confirmed 24-hour urine protein quantity > 1.0g;
  12. Patients with mental disorders who cannot cooperate with treatment;
* Medical history or evidence of disease that may interfere with the test results, prevent participants from participating fully in the study, abnormal treatment or laboratory test values, or other conditions that the investigator considers unsuitable for enrollment. The Investigator considers that there are other potential risks that are not suitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
1 year overall survival rate | 1 year
  The proportion of participants who were alive in the study from treatment to 1 year

SECONDARY OUTCOMES:
overall survival and progression free survival | about 2 years
  The time between the start of treatment and the first progression disease or death (whichever occurs first) from any cause
objective remission rate | about 2 years
  The proportion of total subjects in complete response (CR) and partial response (PR);
Disease control rate | about 2 years
  The proportion of subjects in complete response (CR), partial response (PR) and stable disease (SD) to total subjects;
Duration of remission | about 2 years
  The time between the first partial response or complete response and progression disease or death (whichever occurs first) from any cause
adverse events | about 2 years
  adverse events (AEs) categorized by severity in accordance with the CTC AE Version 5.0

OTHER OUTCOMES:
biomarker | about 2 years
  biomarkers that could potentially predict the therapeutic efficacy of IBI110 and Sintilimab

CONTACTS AND LOCATIONS:
Locations (1):
- Feng Wang, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided